CLINICAL TRIAL: NCT02387073
Title: The Efficacy of Electrical Version of Patient Reported Outcome: Patient Survey
Brief Title: The Efficacy of Electrical Version of Patient Reported Outcome
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: SK Telecom Consortium (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, Professor, Seoul National University Hospital
Other Study IDs: E-PRO; H-1207-088-418 (Other: Seouo National University Hospital)
Record Dates: First submitted 2013-11-29; First posted 2015-03-12 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Spinal Disease
Keywords: outcome assessment; self-reported; patient; clinical outcome
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Electrical version: Electrical version patient reported outcome questionnaire was used for patients who had filled-up same questionnaire in a paper version
  Interventions: Other: Electrical version patient reported outcome questionnaire

INTERVENTIONS:
Other: Electrical version patient reported outcome questionnaire — Assess satisfaction of patients with "electrical version patient reported outcome questionnaire".
  Other Names: Electrical patient reported outcome

SUMMARY:
Recently the importance of electrical PRO system is increased for the accuracy, convenience, and efficiency for both patients and physicians. For the evaluation of quality of life, various self-reported questionnaires is filled-out by the patient, mostly in front of outpatient clinic, and doctor usually take times to calculate the score. If there is electrical PRO which is available with mobile device, the efficacy of clinic would be improved. The investigators developed such a system and applied the system for patients with spinal disease. The investigators assessed the effectiveness of application of electrical-PRO in outpatients' clinic for patients who had filled-up same questionnaire in paper version.

DETAILED DESCRIPTION:
Age, sex, education levels, use of smartphone, the number of applications.

ELIGIBILITY:
Inclusion Criteria:

* We assessed the effectiveness of application of electrical-PRO in outpatients' clinic for patients who had filled-up same questionnaire in paper version

Exclusion Criteria:

* Computer illiterate
* Uncooperative patient

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the patients who have experienced paper questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The necessity of electrical PRO system (quantitative analysis) | up to 6 months after introduction of e-PRO system
  Do you feel the e-PRO system is necessary?
  1. Absolutely yes
  2. Yes
  3. No
  4. Absolutely no

SECONDARY OUTCOMES:
Consultation efficacy with doctor Satisfaction for the enough exchange of information | up to 6 months after introduction of e-PRO system
  Do you feel the e-PRO system make the consultation time with doctor to be efficient?
  1. Absolutely yes
  2. Yes
  3. No
  4. Absolutely no
  Do you think your status was expressed better with the use of e-PRO
  1. Absolutely yes
  2. Yes
  3. No
  4. Absolutely no

CONTACTS AND LOCATIONS:
Overall Officials: Chun Kee Chung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea